CLINICAL TRIAL: NCT06547489
Title: A Phase 2, Multicenter, Randomized, Double-blind Evaluation of the Efficacy and Safety of Oral GATE-251 or Placebo for the Reduction of Symptoms of Major Depressive Disorder in Adults
Brief Title: GATE-251 or Placebo for the Reduction of Symptoms of Major Depressive Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Syndeio Biosciences, Inc (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GATE-251-C-202
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder
Keywords: zelquistinel; GATE-251
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: double-blind, placebo-controlled, fixed dose, parallel groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators and site staff, and outcomes assessors will be blind to treatment with GATE-251 or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GATE-251 (zelquistinel) (Experimental): GATE-251 (zelquistinel) will be administered as a single 10 mg oral tablet one time each week for 6 weeks.
  Interventions: Drug: Zelquistinel
- Placebo (Placebo Comparator): Placebo tablet identical in appearance to the experimental treatment tablet, administered as as a single oral tablet one time each week for 6 weeks.
  Interventions: Drug: Zelquistinel

INTERVENTIONS:
Drug: Zelquistinel — Zelquistinel is a positive allosteric modulator of the N-Methyl-D-Aspartate (NMDA) receptor
  Other Names: GATE-251

SUMMARY:
The goal of this clinical trial is to learn if GATE-251 works to treat depression in adults. It will also learn about the safety of GATE-251. The main questions it aims to answer are:

Does GATE-251 reduce depression scores in participants compared to participants who take a placebo (a look-alike tablet that contains no GATE-251)?

What medical problems are observed in participants who take GATE-251?

Participants will take one tablet of GATE-251 or placebo every week for 6 weeks. Participants will visit the clinic every week of the 6 week period to have the severity of their depression evaluated.

DETAILED DESCRIPTION:
This is a Phase 2 multicenter, randomized, double-blind, placebo-controlled, parallel-group, fixed dose clinical trial designed to evaluate the safety and efficacy of GATE-251 versus placebo in subjects with symptoms of major depressive disorder. Each subject will participate in this study up to 98 days: up to 28 days for screening, 42 days for double-blind treatment, and a 4-week follow-up period. Subjects will return to the clinic one time each week to have the severity of their depression assessed using the Hamilton depression rating scale-17. Adverse events that occurred since the last study visit will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following inclusion criteria to be eligible to participate in the study:

1. Male or female subjects.
2. Aged 18 to 64 years, inclusive.
3. Subject has a diagnosis of major depressive disorder (MDD), single or recurrent episode, defined by the Diagnosis and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5); if single episode, the duration must be ≥3 weeks and ≤18 months. The diagnosis of MDD will be made by a site psychiatrist and supported by the Structured Clinical Interview for DSM-5 - Clinical Trials version (SCID-5-CT) and confirmed by remote, independent raters from the Massachusetts General Hospital Clinical Trials Network and Institute with a State versus trait, Assessability, Face validity, Ecological validity, and Rule of three Ps (pervasive, persistent, and pathological) (SAFER) interview:

   1. The current depressive episode is ≥3 weeks and ≤18 months in duration prior to the Screening Visit (V1);
   2. Have an appropriate severity of illness of at least moderately ill corresponding to a CGI-S score of ≥4 at the Screening and Baseline Visits (V1 and V2, respectively); and
   3. Importantly, have a sufficient history and/or independent report verifying that the current depressive episode is causing clinically significant distress or impairment in functioning.
4. Subject has a Hamilton Depression Rating Scale-17 (HDRS-17) using the Structured Interview Guide for the Hamilton Rating Scale for Depression (SIGH-D) total score of ≥22 at the Screening Visit (V1) and Baseline Visit (V2) with no more than a 25% change from the Screening Visit (V1) to the Baseline Visit (V2).
5. Subject has Hamilton Anxiety Rating Scale (HARS) total score ≥15 at the Screening Visit (V1) and predose at the Baseline Visit (V2).
6. Subject has Insomnia Severity Index (ISI) total score ≥15 at the Screening Visit (V1) and predose at the Baseline Visit (V2)
7. Female subjects must meet 1 of the following:

   1. Surgically sterile or at least 2 years menopausal (ie, postmenopausal is defined as a woman with the absence of menses for at least 12 consecutive months). Menopausal status is to be confirmed by assessing the follicle stimulating hormone level at Screening Visit (V1), or,
   2. If a woman of child bearing potential, subject must use an acceptable method of birth control from date of Screening to the last evaluation at Day 71. Must have a documented negative point of care urine pregnancy test within 24 hours prior to first dosing.
8. Male subjects, including those who are surgically sterile, must use a medically acceptable form of contraception from the time of randomization until the last evaluation at Day 71. Male subjects are strongly advised to inform female partners of the need for them to use highly effective birth control during this time period.
9. Subject must be medically stable by physical examination, medical history, vital signs, laboratory evaluations, and 12-lead electrocardiogram performed at the Screening Visit (V1) and Baseline (V2). If abnormalities are found, the subject may be included if the Investigator, contract research organization (CRO) and sponsor medical monitors judge the abnormalities to be not clinically significant.
10. Ability to understand the nature and requirements of the study and is willing to comply with the study restrictions and agree to return for the required assessments.
11. Provides written informed consent to participate in the trial.
12. Is able to communicate with investigational site personnel, able to complete patient-reported outcome measures and in the opinion of the Investigator, can be reliably rated on assessment scales

Exclusion Criteria:

Any subject who meets any of the following criteria will be excluded from study participation:

1. Evidence of treatment-resistant MDD, defined by having an inadequate response (≤25%) to 2 or more different medications approved for the treatment of MDD at an adequate dose (per locally approved label) for an adequate duration during the current episode using the Massachusetts General Hospital Antidepressant Treatment Rating Questionnaire (ATRQ).
2. Current DSM-5 diagnosis of bipolar (or related disorders), antisocial personality disorder, obsessive compulsive disorder, borderline personality disorder, or attention-deficit/hyperactivity disorder. Subjects not meeting full DSM-5 criteria for borderline personality disorder but exhibiting recurrent suicidal gestures, threats, or self-mutilating behaviors should also be excluded.
3. Subject has a current or prior DSM-5 diagnosis of a psychotic disorder, or MDD with psychotic features.
4. Current concomitant treatment with Food and Drug Administration (FDA)-approved antidepressants, antipsychotics, mood stabilizers, sedatives, or stimulants. Current or past treatment with esketamine, ketamine, or psychedelics is prohibited. Subject must have current concomitant treatment discontinued at least 14 days prior to the Baseline Visit (V2). Subjects may continue anxiolytic agents, except for drugs that are also used to treat depression, or benzodiazepines, or sleep aids [see Section 5.5.1 for a nonexhaustive list] (except trazodone) so long as they have been on a stable dose for at least 3 months and do not intend to change dose during double-blind treatment period (Day 1, Week 1 through end of Week 6 [Day 43]). Subjects who use cannabis or cannabis-derived molecules, including tetrahydrocannabinol (THC), whether natural or chemically-synthesized, hemp seed oil, or cannabidiol (CBD) products (eg, gummies), must be discontinued for at least 14 days prior to the Baseline Visit (V2).
5. Treatment with any experimental antidepressant agent or treatment with a psychedelic agent in an FDA-approved clinical study within the past 12 months.
6. History of electroconvulsive therapy, vagus nerve stimulation, deep brain stimulation, or repetitive transcranial magnetic stimulation within the past 5 years or has had a failure of response to electroconvulsive therapy at any time.
7. Subject has clinically significant renal dysfunction as assessed by the estimated glomerular filtration rate <70 mL/min using the Chronic Kidney Disease Epidemiology Collaboration - creatinine (CKD-EPI creatinine) methodology.
8. Subject has liver protein and enzyme (alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transferase, total bilirubin, lactate dehydrogenase test result >1.5 times the upper limit of normal (subjects with a diagnosis of Gilbert's Syndrome may be eligible if no liver function or enzyme test results other than total bilirubin are >1.5 times upper limit of normal).
9. Subject has resting heart rate (supine) <60 or >100 bpm at the Screening Visit (V1) or predose Baseline (V2).
10. Subject has resting diastolic blood pressure <50 mmHg at the Screening Visit (V1) or predose Baseline (V2).
11. Subject has cardiac PR interval >250 msec at the Screening Visit (V1) or predose Baseline (V2), or QTcF or QTcB interval >450 msec in males or >470 msec in females, or QRS interval >120 msec.
12. Evidence of alcohol abuse (>4 units of alcohol on most days; 1 unit=½ pint of beer, 1 glass of wine, or 1 ounce of hard liquor/spirits) or a positive saliva alcohol screen at Screening (V1) and predose at the Baseline Visit (V2). Alcohol consumption should be avoided for at least 24 hours prior to Baseline Visit (V2).

    Note: Subject may not be rescreened.
13. Abuse of illicit substances, including psychedelic mushrooms by DSM-5 definition of substance use disorder within the 12 months prior to the Screening Visit (V1). Nicotine- containing products eg cigarettes, cigars, vaping, and pipes must be discontinued for at least 14 days prior to randomization. Positive urine test for any drug of abuse is exclusionary.
14. Positive urine test for any drug of abuse (except cannabis or cannabis-derived molecules such as THC whether natural or chemically-synthesized [see exclusion criterion 4]) with the exception of appropriate use of prescribed barbiturates. Subjects may not be rescreened after failing a drug screen.
15. HIV infection, COVID-19 infection, or active hepatitis B or C, syphilis, or other ongoing infectious disease at the Screening Visit (V1).
16. Has laboratory evidence of hypothyroidism at Screening (V1) as measured by thyroid stimulating hormone (TSH) and reflex free thyroxine (T4). If TSH is abnormal and reflex T4 is normal, the subject may be included.
17. Has current unstable diabetes or glycosylated hemoglobin (HbA1c) >7% at Screening (V1).
18. Currently pregnant, planning to become pregnant during the course of the study, or nursing.
19. Currently working a night shift or may be required to work night shift during the course of this study, from Screening through completion of final polysomnography.
20. Malignancy in the last 5 years, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
21. Subject has received new onset psychotherapy or had a change in the intensity of psychotherapy within 8-weeks prior to the Screening Visit (V1).
22. Currently taking prohibited prescription or over-the-counter medications including herbal therapies (eg, echinacea, ginseng, ginko, elderberry, turmeric, ginger, valerian, chamomile, or St John's wort) and THC or cannabis-containing products [see exclusion criteria 4], which may interfere with the required study psychiatric assessments.
23. History of allergy or sensitivity, or intolerance to zelquistinel, NMDAR ligands including ketamine, dextromethorphan, memantine, methadone, dextropropoxyphene, or ketobemidone.
24. Received another investigational drug or device within 90 days of screening in this study.
25. Previously participated in this study or currently enrolled in any other clinical study.
26. Body mass index of >40 kg/m2 at the Screening Visit (V1).
27. Subject is an employee of Worldwide Clinical Trials (hereafter referred to as Worldwide), the Investigator or study site with direct involvement in the study or other studies under the direction of that Investigator or study site, as well as a family member of an employee or of the Investigator, or an employee of Gate Neurosciences, Inc., or a family member of an employee.
28. In the opinion of the Investigator,

    1. The subject has a significant risk for suicidal behavior during the course of participation in the study, or
    2. At the Screening Visit (V1) (the subject scores "Yes" on Items 4 or 5 in the Suicidal Ideation section of the Columbia Suicide Severity Rating Scale (C-SSRS) with reference to a 6-month period prior to Screening Visit (V1), or
    3. At Screening (V1) the subject has had 1 or more suicidal attempts with reference to a 2-year period prior to Screening Visit (V1), or
    4. The subject is considered to be an imminent danger to themself or others, or
    5. At the Baseline Visit (V2) (the subject scores "Yes" on Items 4 or 5 in the Suicidal Ideation section of the C-SSRS
29. The subject is judged by the Investigator or CRO and Sponsor medical monitors to be inappropriate for the study for any reason.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Hamilton Depression Rating Scale-17 (HDRS-17) score compared to placebo | Change in score from baseline 6 weeks
  HDRS-17 is used to assess the severity of depression. The range of scores for the HDRS-17 is 0 - 52 with lower scores indicating a better outcome

SECONDARY OUTCOMES:
Change in the Clinical Global Impressions - Severity (CGI-S) score compared to placebo | Change in score from baseline to 6 weeks
  The CGI-S is a 7-level rating scale used by a clinician to gauge depression severity. The range of scores is 0-7 with lower scores indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Burch, MD, PhD, Study Chair — Gate Neurosciences
Locations (34):
- United States (34):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham-Huntsville, Huntsville, Alabama
  - Wr-Pri, Llc, Encino, California
  - Irvine Clinical Research, Irvine, California
  - CalNeuro Research Group, Los Angeles, California
  - Pacific Clinical Research Management Group LLC, Upland, California
  - Sunwise Clinical Research LLC, Walnut Creek, California
  - MCB Clinical Research Centers, Inc., Colorado Springs, Colorado
  - Mountain View Clinical Research, Denver, Colorado
  - University of Connecticut School of Medicine Psychiatry Department, Farmington, Connecticut
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - D&H Pompano Research Center, LLC, Margate, Florida
  - Premier Clinical Research Institute, Inc., Miami, Florida
  - Miami Dade Medical Research Institute, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - CenExel iRS (iResearch Savannah), Savannah, Georgia
  - Revive Research Institute, Elgin, Illinois
  - KUMC-Wichita, Wichita, Kansas
  - Quantum Research Associates Corp., Louisville, Kentucky
  - Boston Clinical Trials, Boston, Massachusetts
  - Mayflower Clinical, Russells Mills, Massachusetts
  - Vector Clinical Trials, Las Vegas, Nevada
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Insight Clinical Trials LLC, Independence, Ohio
  - Sooner Clinical Research, Inc., Oklahoma City, Oklahoma
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Austin Clinical Trial Partners, Austin, Texas
  - InSite Clinical Research, LLC, DeSoto, Texas
  - Baylor College of Medicine, Psychiatry and Behavioral Sciences, Houston, Texas
  - Clinical Trials of Texas LLC, San Antonio, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Andes Clinical Research, Orem, Utah
  - Northwest Clinical Research Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No